CLINICAL TRIAL: NCT04858061
Title: "ALCO-VR": Virtual Reality Cue Exposure Therapy for the Treatment of Alcohol Use Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Ministry of Health, Spain (Other Government); Ministry of Education and Vocational Training, Spain (Unknown)
Responsible Party: Principal Investigator, Jose Gutierrez Maldonado, Full Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016I078
Record Dates: First submitted 2021-04-12; First posted 2021-04-26 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment-as-usual supplemented with virtual reality cue-exposure therapy (Experimental): Treatment-as-usual supplemented with virtual reality cue-exposure therapy (TAU + VR-CET).
  Interventions: Behavioral: Virtual Reality Cue Exposure Therapy
- Treatment-as-usual (Active Comparator): Only treatment-as-usual (TAU)
  Interventions: Behavioral: Treatment-as-usual

INTERVENTIONS:
Behavioral: Virtual Reality Cue Exposure Therapy — Exposure to alcohol-related cues within virtual environments
  Arms: Treatment-as-usual supplemented with virtual reality cue-exposure therapy
Behavioral: Treatment-as-usual — Pharmacotherapy and psychotherapy
  Arms: Treatment-as-usual

SUMMARY:
Alcohol-related stimuli emerge as high-risk cues for individuals diagnosed with alcohol use disorder (AUD). Relapse after treatment remains a challenge in AUD. Alcohol craving and anxiety are factors contributing to relapse, even after completion of treatment. The current study aims to test the efficacy of a Virtual Reality Cue-Exposure Therapy (VR-CET) patients diagnosed with severe AUD, who made several failed attempts to cease alcohol drinking. It is expected that VR-CET is more efficient in reducing AUD symptomatology and preventing relapses than treatment-as-usual (TAU). 80 participants will be randomly assigned to experimental or control group. The experimental group will receive treatment-as-usual supplemented with 6 sessions of virtual reality cue-exposure therapy (TAU + VR-CET) over the course of five weeks. VR-CET booster sessions consist of exposure to preferred alcoholic beverages and alcohol-related contexts in a VR environment. Throughout the six VR-CET sessions, momentary anxiety and alcohol craving levels will be assessed. The control group will receive only treatment-as-usual (TAU).

DETAILED DESCRIPTION:
The efficacy of VR Cue Exposure Therapy and Cognitive Behavioral Therapy will be investigated on 80 primarly diagnosed by AUD. Participants will be recruited from Hospital Clínico de Barcelona (Barcelona, Spain). They will be randomly assigned to two booster treatments: treatment-as-usual supplemented with 6 sessions of virtual reality cue-exposure therapy (TAU + VR-CET) versus only treatment as-usual (TAU).

Visuo-tactile and visuo-motor stimulation will be induced to participants to get illusory feelings of ownership over the virtual body. Then patients will be choosing their favorite beverages and favorite places to have drinks. During exposure to a specific beverage in VR, participants' olfactory sense will also be stimulated by pouring the beverage onto a cotton and making the participant smell.

* Virtual Reality-based Cue Exposure Therapy (CET-VR): the intervention will consist of 6 sessions (two per week) lasting approximately 50 minutes. Throughout the sessions, the patient will be exposed to an individualized hierarchy of different VR environments that simulate situations and stimuli related to alcohol consumption. During exposure, the level of craving and anxiety experienced by patients will be assessed using visual analog scales. Once the level of craving has decreased sufficiently (40% of the initial level) in a given situation, it will move to another of greater difficulty to complete the hierarchy. The objective of the intervention is to reduce the craving response of patients in these situations through habituation and extinction processes, so that the generalization of the responses learned during treatment to real situations reduces the risk of relapse.
* Treatment-as-usual (TAU): All participants received therapy on an individual and group basis. The primary therapeutic goal of TAU was to maintain abstinence from alcohol during and after treatment discharge. The treatment consisted of a combination of pharmacotherapy and psychotherapy. Pharmacotherapy generally included medication such as disulfiram, anxiolytics, and/or antidepressants. Individual and group therapy sessions were based on psychotherapeutic approaches like cognitive-behavioral therapy and motivational interviewing. Weekly groups included facilitated recovery-oriented discussions in an open-group format. The TAU groups met once or twice weekly for 1 hour and 30 minutes. Patients assigned to the TAU condition were administered two assessment sessions with a 4-5-week diference in-between.

The initial evaluation session will be approximately one hour. The same evaluation instruments with the same procedure will be implemented in the post-treatment session, once finished either virtual reality or cognitive-behavioral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with moderate (4-5 diagnostic criteria) or severe (6 or more diagnostic criteria) AUD according to DSM-5
* Minimum 3 days abstinence before initial evaluation

Exclusion Criteria:

* severe cognitive impairment that could interfere with comprehension and completion of the task
* severe psychopathology (e.g. major depression, schizophrenia, dementia)
* opiate addiction
* epilepsy
* severe visual impairments
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Craving based on AUDIT | pre-assessment
  Change in Craving levels using the Alcohol Use Disorders Identification Test (AUDIT), with scores ranging from 0 to 40. Higher scores reflect higher levels of craving
Change in Craving based on MACS | at pre-assessment and after 3 weeks
  Change in Craving levels using the Multidimensional Alcohol Craving Scale (MACS), with scores ranging from 0 to 60. Higher scores reflect higher levels of craving
Change in Anxiety | at pre-assessment and after 3 weeks
  Change in Anxiety levels using the State-Trait Anxiety Inventory (STAI), with scores ranging from 0 to 60. Higher scores reflect higher levels of anxiety

OTHER OUTCOMES:
Craving levels during exposure sessions | Up to 50 minutes. Baseline (prior to beginning the session), every 20 seconds during the virtual reality session, and at the end of the session
  Visual Analogue Scales from 0-100. Higher scores reflect higher levels of craving
Anxiety levels during exposure sessions | Up to 50 minutes. Baseline (prior to beginning the session), every 20 seconds during the virtual reality session, and at the end of the session
  Visual Analogue Scales from 0-100. Higher scores reflect higher levels of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: José Gutiérrez Maldonado, Prof. Dr., Principal Investigator — University of Barcelona
Locations (1):
- Universitat de Barcelona, Barcelona, Spain